CLINICAL TRIAL: NCT02609607
Title: Treating Anorectal Dysfunction Associated With Multiple Sclerosis
Brief Title: Treating Anorectal Dysfunction in MS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor enrollment; funding ending Dec 31, 2018.
Sponsor: David Levinthal (Other)
Collaborators: Consortium of Multiple Sclerosis Centers (Other)
Responsible Party: Sponsor-Investigator, David Levinthal, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO15100104
Record Dates: First submitted 2015-11-16; First posted 2015-11-20 (Estimated); Results first posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Constipation; Fecal Incontinence; Multiple Sclerosis
MeSH Terms: conditions — Constipation; Fecal Incontinence; Multiple Sclerosis | interventions — Bisacodyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Every other day placement of a placebo rectal suppository for 4 weeks
  Interventions: Other: Placebo
- Bisacodyl (Experimental): Every other day placement of a bisacodyl 10 mg rectal suppository for 4 weeks
  Interventions: Drug: Bisacodyl

INTERVENTIONS:
Drug: Bisacodyl — Rectal suppository
  Other Names: Dulcolax
  Arms: Bisacodyl
Other: Placebo — Rectal suppository
  Arms: Placebo

SUMMARY:
The investigators seek to test whether incorporating the scheduled dosing of a bisacodyl 10 mg rectal suppository every other day improves bowel-related symptoms in patients with multiple sclerosis. Patients will be randomized to receive either a placebo suppository or bisacodyl suppository dosed every other day for 4 weeks.

DETAILED DESCRIPTION:
The majority of patients with multiple sclerosis (MS) suffer from some form of anorectal dysfunction, and these difficulties with bowel function are often ranked as negatively impactful on quality of life as impaired mobility. Despite the significant clinical burden of these symptoms, there remains a paucity of published literature supporting specific therapeutic options to manage anorectal dysfunction in this clinical population. Most bowel regimens rely on either oral laxatives (i.e. PEG-3350) or anti-diarrheal agents (i.e. loperamide). In their study, the investigators propose to establish the efficacy of a bowel regimen that combines both oral agents (as needed; standard care) with scheduled, every other day dosing of a placebo or stimulant laxative rectal suppository -- bisacodyl 10 mg.

Bisacodyl is a stimulant laxative medication that is available over-the-counter. It works by activating nerves in the rectum to elicit rectal contractions which ultimately leading to defecation.

ELIGIBILITY:
Inclusion Criteria:

* MS patients with mild to moderately severe disease (Multiple Sclerosis Impact Scale [MSIS-29] physical domain scores <61 or equivalent Extended Disability Severity Score [EDSS] < 6.5) of any age, gender, disease subtype, duration of illness, current use of MS disease modifying therapy, or comorbid medical condition AND who also have anorectal dysfunction (chronic constipation and/or fecal incontinence) are eligible.

Exclusion Criteria:

* MS patients with severe disease (MSIS-29 physical domain scores greater than 61 or equivalently severe EDSS greater than 6.5), patients with surgically altered anorectal anatomy (i.e. proctectomy/partial colectomy, ostomy creation), active enteric infection (i.e., Clostidium Difficile), or inflammatory bowel disease (i.e. ulcerative proctitis, ulcerative colitis) will also be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-06; Primary Completion 2018-11 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J Levinthal, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Bisacodyl
Started | 6 | 5
Completed | 6 | 4
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Bisacodyl | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 5 | 8
  >=65 years | 3 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (6.3) | 58 (5.2) | 60.6 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 2 | 2 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 30% Improvement From Baseline in Bowel Symptoms at 4 Weeks
Description: All subjects were asked the following question at study entry ('baseline') and the end of 4 weeks of intervention: "Using a scale of 1 to 10 (1 being no problem and 10 being maximally impactful symptoms), how would you rate the severity of your bowel symptoms over the past 2 weeks?"
  The range of reported values was 2-9. We took a response to be a 30% decrease (i.e. improvement) in the subjective symptom score between the baseline and 4 week assessment.
Time Frame: Baseline, 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 6 | 4
Participants | 2 | 0

2. Secondary Outcome: Change From Baseline in Mean PAC-SYM Subscale Scores at 4 Weeks
Description: The Patient Assessment of Constipation Symptom Questionnaire (PAC-SYM) is a validated measure of constipation severity. The questionnaire has a total score and three subscales: Abdominal Symptoms, Rectal Symptoms, and Stool Form. The mean total score and each of the scale subscores are reported in a range of 0-4, with higher scores meaning worse outcomes. A difference (number) of 0.75 in the mean PAC-SYM total and each of the subscale scores is regarded as a clinically significant change.
Time Frame: Baseline, 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 6 | 4
units on a scale
  Change in PAC-SYM Total Score | -0.24 (0.36) | 0.06 (0.49)
  Change in Abdominal Symptoms | 0 (0.16) | 0.13 (0.48)
  Change in Rectal Subscale | 0 (0.76) | -0.42 (0.63)
  Stool Subscale | 0 (1.30) | -0.05 (0.19)

3. Secondary Outcome: Change From Baseline in Fecal Incontinence Severity Index (FISI) Score at 4 Weeks
Description: The Fecal Incontinence Severity Index (FISI) is measures of fecal incontinence severity. The FISI score ranges from 0 to 61, with higher scores interpreted as worse fecal incontinence severity.
Time Frame: Baseline, 4 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 6 | 4
units on a scale | -1.83 (7.9) | 4.25 (19.4)

4. Secondary Outcome: Change From Baseline in Fecal Incontinence Quality of Life (FIQL) Score at 4 Weeks
Description: The Fecal Incontinence Quality of Life (FIQL) Scale measures of the impact of fecal incontinence on aspects of quality of life. There are 4 subscales: Lifestyle, Coping/Behavior, Depression/Self-Perception, and Embarrassment, each of which is calculated as an average score ranging from 1 to 5, with higher scores indicating a greater functional status of quality of life.
Time Frame: Baseline, 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 6 | 4
units on a scale
  Lifestyle | -0.32 (0.41) | -0.1 (0.03)
  Coping / Behavior | -0.22 (0.65) | -0.06 (0.17)
  Depression/ Self-Perception | -0.17 (0.36) | 0.07 (0.21)
  Embarrassment | -0.44 (0.62) | 0.17 (0.69)

5. Secondary Outcome: Change From Baseline in PAC-QOL Scores at 4 Weeks
Description: The Patient Assessment of Constipation Quality of Life (PAC-QOL) Questionnaire is a validated measure of the quality of life impact of constipation. The questionnaire is reported a total score, reported as the average item scores and ranging from 0 to 4, where higher scores represent poorer QOL.
Time Frame: Baseline, 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 6 | 4
units on a scale | -0.04 (0.23) | -0.33 (0.44)

6. Secondary Outcome: Change From Baseline in SF-36 Scores at 4 Weeks
Description: The RAND Health Survey (v.1) is a 36 item questionnaire that measures health in multiple domains. The measure is reported as scores on eight subscales: Physical functioning, Role limitations due to physical health, Role limitations due to emotional problems, Energy/fatigue, Emotional well-being, Social functioning, Pain, and General health. Scores on each subscale range from 0 and 100, with higher scores indicative of better health function in the domain.
Time Frame: Baseline, 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 6 | 4
units on a scale
  Physical functioning | 3.33 (7.45) | -1.25 (5.45)
  Role limitations due to physical health | -16.67 (23.57) | -12.5 (21.65)
  Role limitations due to emotional problems | -7.33 (37.8) | 16.5 (16.5)
  Energy/fatigue | -4.17 (3.44) | -6.25 (7.4)
  Emotional well-being | -5.33 (7.89) | -1 (1.73)
  Social functioning | -4.5 (17.22) | 0 (8.49)
  Pain | 13.67 (19.94) | -1.75 (4.92)
  General health | -4.17 (3.44) | -3.75 (9.60)

7. Secondary Outcome: Change From Baseline In Percent of Subjects With Normal Average Stool Form at 4 Weeks
Description: The Bristol Stool Scale (BSS) is a validated measure of stool form, ranging from 1-7. Normal stool form is regarded as average scores of 3 to 4. Subjects were asked to assess the BSS in their 'bowel diaries' during a preparatory phase of up to 4 weeks prior to study entry and for 4 weeks after intervention, but these 'bowel diaries' were not required for entry into the trial.
Time Frame: Baseline, 4 weeks
Population: Comparative data was available for only 3 of the 6 subjects randomized to placebo, and only 1 of the 4 subjects randomized to receive Bisacodyl.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 3 | 1
percentage of participants | 0 | 0

8. Secondary Outcome: Change From Baseline In Average Number of Daily Bowel Movements at 4 Weeks
Description: Subjects were asked to record each bowel movement in their 'bowel diaries' during a preparatory phase of up to 4 weeks prior to study entry and for 4 weeks after intervention. We used this information to calculate the average difference in number of bowel movements / day before and after exposure to placebo or Bisacodyl. However, these 'bowel diaries' were not required for entry into the trial. Thus, comparative data for bowel movement frequency was available for 3 of the 6 subjects randomized to placebo, and 2 of the 4 subjects randomized to receive Bisacodyl.
Time Frame: Baseline, 4 weeks
Population: These 'bowel diaries' were not required for entry into the trial. Thus, comparative data for bowel movement frequency was available for 3 of the 6 subjects randomized to placebo, and 2 of the 4 subjects randomized to receive Bisacodyl.
Measure: Mean (Standard Deviation); unit: bowel movements per day
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 3 | 2
bowel movements per day | 0.02 (0.70) | -0.21 (0.33)

9. Secondary Outcome: Change From Baseline In Average Number of Fecal Incontinence Episodes at 4 Weeks
Description: Subjects were asked to record each episode of fecal incontinence in their 'bowel diaries' during a preparatory phase of up to 4 weeks prior to study entry and for 4 weeks after intervention. We used this information to calculate the mean difference in the average number of fecal incontinence episodes / day.
Time Frame: Baseline, 4 weeks
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: incontinence episodes per day
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 3 | 2
incontinence episodes per day | 0.05 (0.16) | -0.04 (0.32)

ADVERSE EVENTS:
Time Frame: During trial duration (4 weeks)
Arm/Group | Placebo | Bisacodyl
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6) | Bisacodyl (N=5)
Abdominal cramps (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early Termination due to Difficulty in Recruitment, leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-26): https://cdn.clinicaltrials.gov/large-docs/07/NCT02609607/Prot_SAP_000.pdf